CLINICAL TRIAL: NCT01712503
Title: A Trial of Toric Versus Non-toric Intraocular Lenses in Phacoemulsification Cataract Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Sussex Hospitals NHS Trust (Other)
Collaborators: Rayner Intraocular Lenses Ltd (Unknown)
Responsible Party: Principal Investigator, Mr Masoud Teimory, Consultant ophthalmologist and principle investigator, Western Sussex Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1518/WSHT/2012
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Cataract; Astigmatism
Keywords: Cataract; Astigmatism; Toric; Phacoemulsification; Intraocular lens
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Toric intraocular lens (Experimental): TFlex Lens (623T)
  Interventions: Device: Phacoemulsfication cataract surgery and intra-ocular lens implant
- Monofocal intraocular lens (Placebo Comparator): Superflex Aspheric Lens (920H)/Cflex Aspheric Lens (970C)
  Interventions: Device: Phacoemulsfication cataract surgery and intra-ocular lens implant

INTERVENTIONS:
Device: Phacoemulsfication cataract surgery and intra-ocular lens implant

SUMMARY:
This is a randomised controlled trial that formally compares intra-ocular lenses, which can be used in cataract surgery, one of which is the standard 'monofocal' lens, and the other is the newer toric lens which can correct astgimatism.

The null hypothesis is that both intra-ocular lenses give the same visual outcome in cataract surgery. The alternative hypothesis is that the toric lens, provides a better unaided (without glasses) vision, by correcting the participant's astigmatism.

It has been decided to conduct a randomised controlled trial of the two lenses, as although the toric lenses are endorsed by many case series (which show a reduction in astigmatism), they have not been formally compared to the standard lens. An RCT will enable the formal comparison.

It is expected that this trial will take approximately a year to conduct: six months of recruitment and six months of follow-up. A further six months will be required to analyse the data and prepare a manuscript for publication.

The investigators do not plan to conduct an interim analysis or report as this is a short-trial (six months follow-up) using two alternative lens that are CE marked and already widely used.

Participants who have both cataract and astigmatism will be identified from the GP/optometrist referral letter. They will be seen in specially designated clinics for this research study, which will run alongside the routine cataract 'one' stop clinics at St Richard's Hospital and Worthing Hospital. This will allow for those patients who wish to be part of the study to have all the necessary examination done in one visit and for those who decline participation to be seen in the regular cataract clinic. Potential participants will be sent the research trial information (appendix A) with their appointment letter.

After introducing himself the researcher (who is also a senior cataract surgeon at Western Sussex Hospital Trust), will check if potential participants have had the opportunity to read the trial information that they were sent, or give participants a further copy as required. The key points of the trial will be re-iterated by the researcher and they will be invited to ask any questions about the trialThe researcher will check that the potential participant has read and understood the participant information leaflet. They will answer any questions that the potential participant has and will then take signed consent from those willing to participate.

Only one eye (the 'trial eye') from each patient will be used in the trial. In patients with bilateral cataract, one eye will be selected as the trial eye. This will be the eye that the participant prefers, after consultation with the researcher or surgeon, to have operated first. The participant will be allocated a unique study reference number.

Patients who decline to take part in the trial will be offered cataract surgery as per usual WSHT/NHS procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic cataract for which the patient desires surgery
2. Corneal astigmatism of greater than or equal to 2 dioptres
3. No significant ophthalmic comorbidity

Exclusion criteria

1. <18 years of age
2. Significant ophthalmic co-morbidity
3. Pregnant
4. Medically unfit for cataract surgery
5. Not competent to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Unaided LogMAR visual acuity at 2 months post-operatively

SECONDARY OUTCOMES:
Unaided LogMAR visual acuity at 2 weeks and 6 months post-operatively
Corrected visual acuity at 2 months and 6 months post-operatively
Residual spherical and cylindrical prescriptions at 2 weeks, 2 months and 6 months post-operatively
Patients quality of life questionnaire to assess subjective vision, glare at day/night, subjective colour perception, other symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Sussex Hospital Trust, Worthing and Chichester, West Sussex, United Kingdom